CLINICAL TRIAL: NCT01315977
Title: Orthomolecular Mechanisms of Health Effects of Antioxidant Rich Diets, With Focus on Green Tea (Camellia Sinensis), DNA Protection and Key Biochemical Products/Effects of the Antioxidant Response Element
Brief Title: Dietary Antioxidants, Redox Tone and Health Promotion: an Orthomolecular Study of Interactions
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Our Lady of Maryknoll Hospital (Other)
Responsible Party: Dr Siu-Wai CHOI, Postdoctoral Fellow
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HKCTR-1243
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Antioxidant oxidant balance; Activation of Antioxidant Response Element
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Green tea — Each subject will take either green tea (2%w/v), or water, twice a day for twelve weeks, then wash out for twelve weeks and swap onto the other treatment (either green tea of water) for another twelve weeks in addition to their normal food and beverage intake

SUMMARY:
Aging is associated with increased risk of various diseases, and much attention is given to the use of natural products (like herbs) and 'functional food', such as teas, for healthy aging.

The body is continuously exposed to potentially damaging agents (known as free radicals). The imbalance between the amount of free radicals and that of antioxidants in the body is known as oxidative stress. It is known that Type 2 DM is a state of increased oxidative stress, which is thought to lead to many long term complications of Type 2 DM, such as heart disease, vision problems and kidney failure. Antioxidant therapy, including increased consumption of antioxidant rich foods and beverages such as green tea, has been suggested as possibly beneficial in lowering the risk of these complications.

The purpose of this study is to examine the effects of regular intake of green tea on indices of oxidative stress and antioxidant defense within cells, plasma and urine so as to investigate if regular intake of green tea can be recommended for health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM subjects
* Genotyped for polymorphism in the heme-oxygenase gene promoter region to be homozygous for long (> 26) or short (< 24) GT repeats

Exclusion Criteria:

* smokers
* have suffered DM related complication
* already taking antioxidant or herbal supplements

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Activation of Antioxidant Response Element After Consumption of Green Tea | 12 weeks
  Biomarkers of antioxidant and oxidant balance, antioxidant response element activation (through gene and protein expression studies and plasma biomarkers) will be determined pre and post consumption of green tea

CONTACTS AND LOCATIONS:
Overall Officials: Iris BENZIE, DPhil, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Our Lady of Maryknoll Hospital, Kowloon, Hong Kong, China